CLINICAL TRIAL: NCT01293318
Title: Copeptin Pancreatitis Trial
Brief Title: Study of Copeptin as a Diagnostic Marker for Acute Pancreatitis
Acronym: COPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 281/10
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Acute Pancreatitis; Pancreatitis
Keywords: Copeptin; Vasopressin; antidiuretic hormone (ADH)
MeSH Terms: conditions — Pancreatitis; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute pancreatitis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to investigate if there is an association between copeptin level in serum and the severity of pancreatitis and if copeptin can be used as a predictor for organ failure and pancreatic necrosis with or without superinfection.

DETAILED DESCRIPTION:
Acute pancreatitis may range from mild to severe disease with high mortality in case of infected pancreatic necrosis. Due to its rising incidence it remains an important healthcare problem in Europe and US. The assessment of the severity of pancreatitis is crucial for the further management and the prognosis. Several quite complex scores like Ranson or APACHE II scores has been used in the past with reasonable sensitivity for necrosis or superinfection as well as inflammation markers like c-reactive Protein.

Copeptin, the C-terminal part of antidiuretic hormone, is a relatively stable peptide in blood circulation. Several studies investigated Copeptin in the presence of Systemic Inflammatory Response Syndrome (SIRS) or sepsis, myocardial infarction, lower respiratory tract infection and cerebral stroke. Copeptin has shown to be a helpful prognostic marker in these diseases. The aim of this prospective study is to investigate whether Copeptin can be used to assess the severity of pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pancreatitis
* written informed consent
* inpatient treatment

Exclusion Criteria:

* time interval between onset of abdominal symptoms and study inclusion >96h
* patients unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency departement or in-hospital patients with acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Association between copeptin level and severity of pancreatitis (according to Atlanta classification) | 48 hours
  Copeptin level will be measured on admission into hospital and severity of pancreatitis will be classified according to the Atlanta criteria.

SECONDARY OUTCOMES:
Comparison of copeptin with C reactive protein and procalcitonin in terms of assessing severity of pancreatitis | 48 hours
Predictive accuracy of copeptin, C reactive Protein (CRP) and procalcitonin in terms of developing organ failure, necrosis and/or superinfection and mortality | Duration of hospitalisation
  Determinating Atlanta score, Sofa score. Assessing local complications by checking CT scan and searching for superinfection in fine needle aspiration and/or biopsy.
Determine whether change in copeptin level from day 0 to 2 is associated with organ failure, necrosis and/or superinfection | Duration of hospitalisation
  To determine if the change in copeptin level is associated with organ failure, necrosis and superinfection

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Nebiker, MD, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Morgenthaler NG, Muller B, Struck J, Bergmann A, Redl H, Christ-Crain M. Copeptin, a stable peptide of the arginine vasopressin precursor, is elevated in hemorrhagic and septic shock. Shock. 2007 Aug;28(2):219-26. doi: 10.1097/SHK.0b013e318033e5da. PMID 17515850
- [Background] Muller B, Morgenthaler N, Stolz D, Schuetz P, Muller C, Bingisser R, Bergmann A, Tamm M, Christ-Crain M. Circulating levels of copeptin, a novel biomarker, in lower respiratory tract infections. Eur J Clin Invest. 2007 Feb;37(2):145-52. doi: 10.1111/j.1365-2362.2007.01762.x. PMID 17217381
- [Background] Stolz D, Christ-Crain M, Morgenthaler NG, Leuppi J, Miedinger D, Bingisser R, Muller C, Struck J, Muller B, Tamm M. Copeptin, C-reactive protein, and procalcitonin as prognostic biomarkers in acute exacerbation of COPD. Chest. 2007 Apr;131(4):1058-67. doi: 10.1378/chest.06-2336. PMID 17426210
- [Background] Katan M, Fluri F, Morgenthaler NG, Schuetz P, Zweifel C, Bingisser R, Muller K, Meckel S, Gass A, Kappos L, Steck AJ, Engelter ST, Muller B, Christ-Crain M. Copeptin: a novel, independent prognostic marker in patients with ischemic stroke. Ann Neurol. 2009 Dec;66(6):799-808. doi: 10.1002/ana.21783. PMID 20035506